CLINICAL TRIAL: NCT02032420
Title: A Double Blinded Randomized Controlled Trial on the Effects of Four Sequential Maneuvers on Ultrasound Guided Nerve Block Performance
Brief Title: The Effects of the STAR Maneuver on UGRA Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Timothy R Petersen, Research Information Specialist, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STAR vs. ART
Record Dates: First submitted 2013-12-18; First posted 2014-01-10 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2016-12

CONDITIONS: Simulator-based Training of Ultrasound-guided Regional Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- STAR (Experimental): Introductory training by video depicting 4 sequential maneuvers for reacquisition of needle image in ultrasound: see, tilt, align, rotate.
  Interventions: Behavioral: STAR
- ART (Active Comparator): Introductory training with a video depicting 3 probe position aspects for reacquisition of needle image by ultrasound: alignment, rotation, tilt.
  Interventions: Behavioral: ART

INTERVENTIONS:
Behavioral: STAR
  Arms: STAR
Behavioral: ART
  Arms: ART

SUMMARY:
Volunteers will watch a training video demonstrating how to place a needle in the correct position while keeping it visible. Later the volunteers will be placed in front of a set up identical to the video, and asked to demonstrate how to direct an 80 mm echogenic Pajunk needle into 3 targets in a standardized homemade phantom a total of three times.

DETAILED DESCRIPTION:
After watching the training video, each volunteer will be placed in front of a set up identical to the video seen. Adjacent to this set up, a single fellowship trained regional anesthesiologist known as the assessor is situated with a screen that allows real time viewing of the ultrasound screen seen by the volunteer. The assessor is blinded to the assignment of the volunteer. Also, the assessor does not have any visualization of the volunteer. This prevents visualizing hand or body movement that may cause a bias. The same assessor is used for the whole study to provide consistent assessment of the task.

The task involves the volunteer directing an 80 mm echogenic Pajunk needle into 3 targets in a standardized homemade phantom. The targets simulate the nerve roots commonly found in the interscalene block. Thus, they are arranged diagonally to simulate the nerve root position commonly seen. Also, they are arranged on a tilt relative to the flat surface of the phantom to simulate the direction the nerve travels. This is important as the tilt of the target requires the volunteer to tilt the probe so that their incidental ultrasound wave is perpendicular to the target for the brightest reflection to occur. This phenomenon is known as anisotropy. This increases the realism of the task that cannot be imitated by commercially available phantoms.

There are 3 goals that the volunteer must fulfill in performing their task. Firstly, they must direct the needle to the 12 o'clock position of the 3 targets. Secondly, they must achieve maximal ultrasound image brightness of the 3 targets at all times. Thirdly, the entire needle must be visualized at all times.

If the needle is not in the correct position, the assessor will verbally inform the volunteer to redirect it to the correct position. If the target images are not at their brightest, the assessor will verbally inform the volunteer not to manipulate the needle towards the target until the targets are at their brightest. Clinically, this functions to prevent the needle being inserted inside the nerve as the targets are not clearly seen. Thirdly, if the needle is visualized entirely, the volunteer will be told to stop manipulating the needle towards the target until the needle is fully visualized by manipulating the probe. A timer records the cumulative time the needle is not in full visualization. Clinically, this functions to prevent the needle being inserted into a nerve or structure that it should not.

After all 3 targets have been completed, the volunteer repeats the task a total of 3 times.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Right handed
* Aged 18 to 55

Exclusion Criteria:

* Any person who has prior knowledge about ultrasound imaging or regional anesthesia
* Any person who has prior experience with laparoscopy or biopsy
* Any person who has problems with depth of field or simple hand eye co-ordination task

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Lam, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Hospital, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- STAR Strategy: Introductory training by video depicting 4 sequential maneuvers for reacquisition of needle image in ultrasound: see, tilt, align, rotate.
- ART Strategy: Introductory training with a video depicting 3 probe position aspects for reacquisition of needle image by ultrasound: alignment, rotation, tilt.
Period: Overall Study
Arm/Group | STAR Strategy | ART Strategy
Started | 18 | 17
Completed | 18 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | STAR Strategy | ART Strategy | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 21 [19 to 23.25] | 21 [19 to 23.5] | 21 [19 to 23]
Gender [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 11 | 5 | 16
Plays video games [Number; unit: participants] | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Task Completion Time
Description: Median time taken to complete 3 iterations of the assigned task, across participants within a study arm
Time Frame: Immediately after training
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | STAR Strategy | ART Strategy
Number analyzed (Participants) | 18 | 17
seconds | 87 [47.8 to 116.1] | 343 [214 to 600]
Statistical Analysis 1: Comparison: STAR Strategy vs ART Strategy; Test type: Superiority or Other; p < 0.001, Repeated-measures MANOVA; The reported p value is for the effect of group assignment across three iterations of the assigned task

2. Secondary Outcome: Needle-not-seen Time
Description: Median percentage of attempt time on 3 iterations in which the needle is not adequately visualized, across participants within a study arm
Time Frame: During attempt
Measure: Median (Inter-Quartile Range); unit: percentage of attempt time
Arm/Group | STAR Strategy | ART Strategy
Number analyzed (Participants) | 18 | 17
percentage of attempt time | 42.8 [32.3 to 68.9] | 68.7 [64.6 to 75.1]
Statistical Analysis 1: Comparison: STAR Strategy vs ART Strategy; Test type: Superiority or Other; p = 0.004, Repeated-measures MANOVA; The p value is for the effect of group assignment across three iterations of the assigned task

3. Secondary Outcome: Performer Fatigue
Description: Self-reported trainee fatigue on a numerical rating scale (1= least fatigued; 10=most fatigued); lower scores indicate less fatigue
Time Frame: During task
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | STAR Strategy | ART Strategy
Number analyzed (Participants) | 18 | 17
units on a scale | 1 [1 to 2.5] | 4.5 [1 to 9]
Statistical Analysis 1: Comparison: STAR Strategy vs ART Strategy; Test type: Superiority or Other; p = 0.038, Wilcoxon (Mann-Whitney)

4. Post Hoc Outcome: Inability to Complete Assigned Task at All in Three Attempts
Description: Some participants found the task too difficult to complete.
Time Frame: Immediately after training
Measure: Number; unit: participants
Arm/Group | STAR Strategy | ART Strategy
Number analyzed (Participants) | 18 | 17
participants | 0 | 7
Statistical Analysis 1: Comparison: STAR Strategy vs ART Strategy; Test type: Superiority or Other; p = 0.003, Fisher Exact

ADVERSE EVENTS:
Time Frame: Immediately after completion of training and assigned tasks
Arm/Group | STAR Strategy | ART Strategy
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No